CLINICAL TRIAL: NCT01975285
Title: Prospective Randomized Double Blind Study to Evaluate the Efficacy of Popliteal Nerve Blocks With and Without Dexamethasone on the Duration of Analgesia for Foot & Ankle Surgery.
Brief Title: Efficacy of Popliteal Nerve Blocks With and Without Dexamethasone on the Duration of Analgesia for Foot & Ankle Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Residency program director, Department of anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00032547
Record Dates: First submitted 2013-10-29; First posted 2013-11-04 (Estimated); Results first posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-04

CONDITIONS: Foot and Ankle Procedures
Keywords: Pain management; Postoperative opioid requirements; Perioperative outcomes; Dexamethasone; Anesthetic adjuvant; Analgesic adjuvant
MeSH Terms: conditions — Agnosia | interventions — Dexamethasone; Calcium Dobesilate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone group (Active Comparator): Dexamethasone 4mg(1 ml) per 20cc
  Interventions: Drug: Dexamethasone
- Saline group (Placebo Comparator): Saline 1 ml per 20cc
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — 0.5% Bupivacaine with 1:200,000 epinephrine + Dexamethasone 4mg per 20cc
  Other Names: Decadron
  Arms: Dexamethasone group
Drug: Saline — 0.5% Bupivacaine with 1:200,000epinephrine + Saline 1 ml per 20cc
  Other Names: placebo
  Arms: Saline group

SUMMARY:
The purpose of this research study to evaluate the effects of dexamethasone as an addition to peripheral nerve block (Put the nerve to sleep with Bupivacaine a numbing medication) on length of pain relief (analgesia), postoperative narcotic (opioids) requirements, pain scores, and patient satisfaction after foot and ankle procedures.

ELIGIBILITY:
Inclusion Criteria:

* 60 patients (30 per group) undergoing foot and ankle procedures
* Willingness and ability to sign an informed consent document
* No allergies to anesthetic or analgesic medications
* American Society of Anesthesiologists (ASA)physical status Class I - III
* Aged 18-90 years,either sex

Exclusion Criteria:

* Refusal to participate in the study
* Age<18 or> 90 years -
* Contraindications to regional blockage including but not limited to:
* Patient refusal to regional blockade
* Infection at the site of needle insertion
* Systemic infection
* Bleeding diathesis or coagulopathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone Group: 0.5% Bupivacaine with 1:200,000epinephrine + Dexamethasone 4mg(1 ml) per 20cc
  Dexamethasone: 0.5% Bupivacaine with 1:200,000 epinephrine + Dexamethasone 4mg per 20cc
- Saline Group: 0.5% Bupivacaine with 1:200,000epinephrine + Saline 1 ml per 20cc
  Saline: 0.5% Bupivacaine with 1:200,000epinephrine + Saline 1 ml per 20cc
Period: Overall Study
Arm/Group | Dexamethasone Group | Saline Group
Started | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 2
Not completed — Failed Block and follow up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Group | Saline Group | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (15) | 55 (14) | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 19 | 17 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 25 | 25 | 50
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: Postoperative pain will be measured using a Verbal Rating Scale (0-10) Verbal Rating Scale: 0 to 10 scale where 0 indicates= No pain" and 10 indicates= The worst possible pain
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dexamethasone Group | Saline Group
Number analyzed (Participants) | 28 | 28
Scores on a scale | 0.21 (0.56) | 0.05 (0.22)

2. Secondary Outcome: Opioid Consumption
Description: Opioid consumption obtained from the recorded data Perioperative use of opioid consumption inside hospital (recorded by study staff and data obtained from patient charts)
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Opioids consumption mg
Arm/Group | Dexamethasone Group | Saline Group
Number analyzed (Participants) | 28 | 28
Opioids consumption mg | 0 (0) | 0 (0)

3. Secondary Outcome: Length of Analgesia
Description: Time in days and/or hours
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Dexamethasone Group | Saline Group
Number analyzed (Participants) | 28 | 28
Hours | 36 [25 to 51] | 30 [22.5 to 41.5]

4. Secondary Outcome: Patient Satisfaction With Regional Nerve Block
Description: Patient satisfaction with regional nerve block: measured using a Verbal Rating Scale (0-10) Verbal Rating Scale: 0 to 10 scale where 0 indicates= No satisfied at all 10 indicates= Extremely satisfied
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dexamethasone Group | Saline Group
Number analyzed (Participants) | 28 | 28
Scores on a scale | 9.6 (0.9) | 9.3 (1.8)

5. Secondary Outcome: Patient Satisfaction With Pain Management
Description: Patient satisfaction with pain management: measured using a Verbal Rating Scale (0-10) Verbal Rating Scale: 0 to 10 scale where 0 indicates= No satisfied at all 10 indicates= Extremely satisfied
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dexamethasone Group | Saline Group
Number analyzed (Participants) | 28 | 28
Scores on a scale | 9 (1.7) | 9.3 (1.4)

ADVERSE EVENTS:
Arm/Group | Dexamethasone Group | Saline Group
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No